CLINICAL TRIAL: NCT06971523
Title: A Multi-center, Open-label, Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of CTS3497 in Patients With MTAP Deficient Advanced Solid Tumors and Lymphomas
Brief Title: A Phase I/II Clinical Study of CTS3497 in Patients With MTAP Deficient Malignacies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CytosinLab Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTS3497-CI01
Record Dates: First submitted 2025-04-28; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor; Lymphoma
Keywords: PRMT5
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I: CTS3497 Monotherapy Dose Escalation/Dose Expansion (Experimental): 7 dose groups are pre-specified in Dose Escalation,and 2-3 dose groups in Dose Expansion.
  Interventions: Drug: CTS3497
- Phase II: CTS3497 Monotherapy Expansion (Experimental): CTS3497 RP2D administered to patients with MTAP homozygous deletion including the following cohorts: esophageal squamous cell carcinoma [ESCC], pancreatic adenocarcinoma [PAAD], biliary tract cancer [BTC], non-small cell lung carcinoma[NSCLC], malignant pleural mesothelioma [MPM], Urothelial cancer, high-grade gliomas, other solid tumors, and lymphomas.
  Interventions: Drug: CTS3497

INTERVENTIONS:
Drug: CTS3497 — CTS3497: Orally via capsules
  Other Names: CTS3497 capsules

SUMMARY:
The primary objective of Phase I of this study is to evaluate the safety and tolerability, and to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of CTS3497 in patients with metastatic or locally advanced methylthioadenosine phosphorylase (MTAP)-deficient solid tumors and lymphomas.

The primary objective of Phase II of this study is to evaluate the efficacy of CTS3497 in patients with metastatic or locally advanced MTAP-deficient solid tumors and lymphomas.

DETAILED DESCRIPTION:
The primary objective of Phase I of this study is to evaluate the safety, tolerability, PK, PD and efficacy to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of CTS3497 in patients with metastatic or locally advanced methylthioadenosine phosphorylase (MTAP)-deficient solid tumors and lymphomas.

The primary objective of Phase II of this study is to evaluate the efficacy and safety of CTS3497 in patients with metastatic or locally advanced MTAP-deficient solid tumors and lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the signing of ICF.
* Patients with histologically or cytologically confirmed locally advanced or metastatic solid tumors who cannot be treated surgically and have failed standard of care (SoC). Or patients with refractory/relapsed lymphomas.
* MTAP deficiency is confirmed by IHC or NGS.
* At least one evaluable tumor lesion at screening for patients in escalation part, and at least one measurable tumor lesion for patients in expansion part.
* ECOG performance status of 0 to 1.
* Adequate hematopoietic function, cardiac function, liver function, renal function, and coagulation function per local laboratory.

Exclusion Criteria:

* Female patients in pregnancy or lactation.
* Patients with dysphagia; or a condition that seriously affects gastrointestinal absorption.
* Allergic or intolerant to the active ingredients or excipients of the investigational product.
* Anti-tumor therapy within 28 days of study day 1.
* Prior treatment with an methionine adenosyltransferase 2α (MAT2A) inhibitor or a protein arginine methyltransferase 5 (PRMT5) inhibitor.
* Central nervous system (CNS) metastasis at screening.
* Live vaccine therapy within 4 weeks before study drug administration.
* Use of therapeutic anti-coagulation for treatment of active thromboembolic events.
* Use of prescription medications that are known strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A4) within 14 days or 5 half-lives (whichever is longer) before study day 1.
* Unresolved toxicity from prior anti-cancer therapy.
* Active infection of HIV, HBV or HCV.
* Patients who are judged by the investigator to have a history of other serious systemic diseases, or not suitable for participating in the trial for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: Number of Patients Who Experience a Dose-Limiting Toxicity (DLT) | Up to 21 days after the first administration.
  Incidence of DLT(s) during the DLT observation period
Phase I: Number of Patients Who Experience a Treatment-emergent Adverse Event (TEAE) | Baseline through 28 days after the end of treatment, estimated up to 52 weeks.
  Adverse events (AEs) are defined as any untoward medical occurrence in clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are any event that occurs after the participant has received study treatment. Any clinically significant changes in vital signs, electrocardiograms (ECGs) and clinical laboratory tests will be recorded as TEAEs.
  Serious AEs (SAEs) are defined as any event that meets at least 1 of the following criteria:
  resulting in death (fatal); requiring in-patient hospitalization or prolongation of existing hospitalization; resulting in persistent or significant disability/incapacity; being a congenital anomaly/birth defect; other medically important serious event.
Phase II: Objective Response Rate (ORR) | up to 48 weeks.
  The percentage of participants having complete response (CR) or partial response (PR) assessed based on RECIST V1.1.

SECONDARY OUTCOMES:
Cmax of CTS3497 | Cycle 1 (each cycle is 21 days) Day 1, Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 5 Day 1
  Maximal Plasma Concentration
Tmax of CTS3497 | Cycle 1 (each cycle is 21 days) Day 1, Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 5 Day 1
  Time to Achieve Maximal Plasma Concentration
AUC of CTS3497 | Cycle 1 (each cycle is 21 days) Day 1, Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 5 Day 1
  Area Under the Plasma Concentration Versus Time Curve
Disease control rate (DCR) | up to 48 weeks.
  Disease Control Rate assessed by investigators based on RECIST v1.1
Duration of Response (DoR) | Estimated up to 48 weeks.
  Duration of response (DOR) assessed based on the Response Evaluation Criteria in Solid Tumors (RECIST) V1.1.
Progression-Free Survival (PFS) | Estimated up to 48 weeks.
  Progression-Free Survival assessed by investigators based RECIST v1.1
Overall Survival (OS) | Up to approximately 3 years.
  Overall Survival after first dose
Pharmacodynamic (PD) characteristics of CTS3497: symmetric dimethylarginine (SDMA) | Cycle 1 (each cycle is 21 days) Day 1, Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 5 Day 1 and Cycle 7 Day 1
  To explore the changes of symmetric dimethylarginine (SDMA) in blood of patients with solid tumors and lymphomas before and after administration of CTS3497.
Pharmacodynamic (PD) characteristics and efficacy analysis. | Estimated up to 48 weeks.
  The correlation between the changes of symmetric dimethylarginine (SDMA) in blood of patients and the efficacy of CTS3497

CONTACTS AND LOCATIONS:
Overall Officials: Haiping Wu, PhD, Study Chair — CytosinLab Therapeutics Co., Ltd.
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China